CLINICAL TRIAL: NCT04026061
Title: Randomised Controlled Feasibility Study Into FindMyApps; First Evaluation of a Tablet Intervention to Promote Self-management and Meaningful Activities in People With Mild Dementia
Brief Title: Pilot Study Person-centred Tablet Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saxion University of Applied Sciences (Other)
Collaborators: University of Twente (Other); Radboud University Medical Center (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FindMyApps
Record Dates: First submitted 2019-07-09; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Dementia; Mobile Applications; Computers; Neurological Rehabilitation; Activities of Daily Living
Keywords: Medical Research Framework; Hand-held touchscreen devices; Self-management; Meaningful activities
MeSH Terms: conditions — Dementia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMA group (Experimental): Receiving the FMA training and tool
  Interventions: Behavioral: FMA group
- control group (Placebo Comparator): Receiving a simple tablet training and some websites
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: FMA group — A person-centred, tailored tablet intervention, called FindMyApps (FMA). The intervention consists of the FMA training to use the tablet and the FMA selection tool to help users find apps for self-management and meaningful activities that fit their needs, wishes and abilities
  Arms: FMA group
Behavioral: Control group — Receiving an introductory tablet training and some links to websites that recommend usable apps for people with dementia in general
  Arms: control group

SUMMARY:
First evaluation of FindMyApps, a tablet intervention consisting of a selection tool for usable apps for self-management and meaningful activities and a training that supports informal carers to help people with dementia to learn how to use the tablet and the tool.

DETAILED DESCRIPTION:
Testing the feasibility and mechanism of impact of FindMyApps, a tablet intervention consisting of a selection tool to help persons with dementia find usable apps for self-management and meaningful activities and a training that supports informal carers to employ errorless learning principles to help people with dementia to learn how to use the tablet and the tool.

An exploratory pilot randomized controlled trial was carried out with a mixed-methods design. Twenty persons with mild dementia and carer dyads were randomly assigned to the FindMyApps group (n = 10) that used the FindMyApps training and selection tool, or a control condition that just got a tablet (n = 10). After informal carers had received the training, the dyads in the experimental group started with the three-month intervention. Pre and post-test measurements consisted of questionnaires and post-test semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Eligible dyads had to be community dwelling.
* Persons with dementia had Mild Cognitive Impairment or mild dementia with a score of 3 to 4 on the Global Deterioration Scale (GDS; 45), with or without a confirmed diagnosis.
* Availability of an informal carer or volunteer to provide support.

Exclusion Criteria:

* Participation in another intervention trial
* Severe visual and/or physical impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Self-management abilities people with dementia | At baseline and post-intervention at 3 months follow up
  Measured with the revised 30-item Self-Management Ability Scale (SMAS-30). Change/ difference between baseline and post-intervention. It consists of six subscales: Taking Initiative, Self-efficacy, Investing, Positive Perspective, Multifunctionality, and Variety. Each subscale consists of five items scored on a 5-point or 6-point Likert-type scale. A 5-point scale is used for 'Self-efficacy' (1 = I certainly do not think so, 5 = I certainly think so) and 'Positive Perspective' (1 = No!, 5 = Yes!), and a 6-point scale is used for 'Taking Initiative', 'Investing', and 'Multifunctionality' (1 = never, 6 = very often), and 'Variety' (1 = none, 6 = more than six). Item scores are transformed into scores ranging from 0 to 20. Mean subscale scores range from 0 to 100, as does the total score, which is the mean score of the six subscales. A higher score indicates more self-management abilities.
Participation in daily and social activities people with dementia | At baseline and post-intervention at 3 months follow up
  Measured with a short version of the Pleasant Activities List (PAL). Change/ difference between baseline and post-intervention. The PAL was used to assess the frequency and enjoyability of daily and social activities. In this study, the PAL was shortened from its original 139 item to 31 items divided into two subscales: Social Activities (SA), such as visiting family, and Domestic Activities (DA), such as gardening. Shortening was done for two reasons: the length of the original version was thought to be not feasible for the PwDs and a focus on social and domestic activities was more in line with this study. Items relate to the frequency of engagement and the subjective enjoyability, which are scored on a 5-point Likert-type scale ranging from 1 (not at all) to 5 (very much). A higher score indicates that activities are done more often and enjoyed more.
Participation in daily and social activities people with dementia | At baseline and post-intervention at 3 months follow up
  Measured with one item of the Adult Social Care Outcomes Toolkit (ASCOT). Change/ difference between baseline and post-intervention. Responses on this item are given on a scale ranging from 1 ('I have as much social contact as I want with people I like') to 4 ('I have little social contact with people and feel socially isolated'). A higher score indicates less social participation.
Feeling of competence informal carers | At baseline and post-intervention at 3 months follow up
  Measured with the Short Sense of Competence Scale (SSCQ). Change/ difference between baseline and post-intervention.The SSCQ contains of seven statements. Informal caregivers had answered these questions on a 5-point-likert scale which ranges from 'agree very strongly' to 'disagree very strongly'. For feeling of competence, the scores on all items were summed to get a sum-score. The sum-score ranges between 7 and 35 and a higher score indicates a greater feeling of competence.

SECONDARY OUTCOMES:
Perceived self-efficacy people with dementia | At baseline and post-intervention at 3 months follow up
  Measured with the Dutch version of the 10-item General Self-Efficacy Scale (D-GSE scale). Change/ difference between baseline and post-intervention. Responses are structured on a 4-point scale ranging from 1 (not at all true) to 4 (exactly true). A total score ranging between 10 and 40 is obtained by summing the responses on all ten items; a higher score indicates more self-efficacy.
Perceived autonomy people with dementia | At baseline and post-intervention at 3 months follow up
  Measured with the 12-item Experienced Autonomy List (EAL). Change/ difference between baseline and post-intervention. Responses are scored on a 5-point Likert scale ranging from 1 (totally disagree) to 5 (totally agree). Responses to negatively worded items are reverse-coded. The scores on all items were summed to get a sum-score. The sum-score ranges between 12 and 60. A higher score indicates more perceived autonomy.
Quality of life people with dementia | At baseline and post-intervention at 3 months follow up
  Measured with the Dementia Quality of Life scale (DQoL). Change/ difference between baseline and post-intervention. It consists of 29 items that are focused on five domains: self-esteem, positive affect, negative affect, feelings of belonging, and sense of aesthetics. All items are rated on a 5-point Likert-type scale. Responses on 'sense of aesthetics' relate to enjoyment and range from 1 (not at all) to 5 (a lot). Responses on the four other subscales relate to frequency and range from 1 (never) to 5 (very often). Scores for the subscales are calculated by computing the mean score. In addition, the DQoL contains one global item to assess overall quality of life on a scale from 1 (bad) to 5 (excellent). A higher score on both the subscales and the global item indicates a higher quality of life.
Positive care experiences informal carers | At baseline and post-intervention at 3 months follow up
  Measured with the Positive Experience Scale (PES). Change/ difference between baseline and post-intervention. The PES is an 8-item scale. The answer categories were: (1) agree , not agree/not disagree and disagree, whereby not agree/not disagree are took together as (0) disagree. The scores on all items were summed to get a sum-score. The sum-score ranges between 0 and 8, whereby a higher score indicates more positive care experiences.
Quality of life informal carers | At baseline and post-intervention at 3 months follow up
  Measured with the EuroQol-5 Dimensions-5 Levels scale (EQ-5D-5L). Change/ difference between baseline and post-intervention. The EQ-5D-5L consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Informal caregivers had the following answer options on these dimensions: (1) no problems, (2) slight problems, (3) moderate problems, (4) severe problems or (5) extreme problems. A mean sum-score was calculated on these dimensions which ranges from 1 till 5, whereby a higher score indicates more problems. Besides that, the EQ-5D-5L consists of the EuroQol Vertical Visual Analogue Scale (EQ VAS), which contains of a 20 centimeter vertical scale ranging from 0 till 100. Informal caregivers rated their health on this scale, whereby a higher score indicates a better health.
Quality of life informal carers | At baseline and post-intervention at 3 months follow up
  Measured with The Older Persons and Informal Caregivers Survey Minimum DataSet (TOPICS-MDS). Change/ difference between baseline and post-intervention. In the quality of life topic of TOPICS-MDS informal caregivers were asked to rate their current quality of life on a five-level response scale which ranges from 1 (excellent) till 5 (poor). Besides that, informal carers rated their quality of life in comparison with the previous year on a five-level response scale which ranges from to 1 (much better) till 5 (much worse), whereby a lower score indicates a better quality of life. The last question which informal caregivers answered was about their perceived quality of life. Informal carers answered this question by rating their present life on a scale of 0 till 10, whereby a higher score indicates a better life.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Kerkhof, MSc, Principal Investigator — Saxion University of Applied Sciences
Locations (1):
- Saxion University of applied Sciences, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerkhof Y, Pelgrum-Keurhorst M, Mangiaracina F, Bergsma A, Vrauwdeunt G, Graff M, Droes RM. User-participatory development of FindMyApps; a tool to help people with mild dementia find supportive apps for self-management and meaningful activities. Digit Health. 2019 Mar 26;5:2055207618822942. doi: 10.1177/2055207618822942. eCollection 2019 Jan-Dec. PMID 30944726
- [Background] Kerkhof YJ, Graff MJ, Bergsma A, de Vocht HH, Droes RM. Better self-management and meaningful activities thanks to tablets? Development of a person-centered program to support people with mild dementia and their carers through use of hand-held touch screen devices. Int Psychogeriatr. 2016 Nov;28(11):1917-1929. doi: 10.1017/S1041610216001071. Epub 2016 Jul 18. PMID 27425002
- [Background] Kerkhof Y, Bergsma A, Graff M, Droes RM. Selecting apps for people with mild dementia: Identifying user requirements for apps enabling meaningful activities and self-management. J Rehabil Assist Technol Eng. 2017 Jun 2;4:2055668317710593. doi: 10.1177/2055668317710593. eCollection 2017 Jan-Dec. PMID 31186930
- See also: Information and enrollment site for future study FMA — http://findmyapps.onderzoek.io/